CLINICAL TRIAL: NCT03464890
Title: Soothing and Re-epithelizing Activity of New Cosmetic Formulations in Comparison to Placebo and Untreated Control Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Medical Doctor, Derming SRL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2017
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Sensitive Skin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LICHTENA DermAD (Experimental): Comparison within subjects of "P926 - LICHTENA DermAD CREMA VISO" and "P927 - LICHTENA DermAD CREMA CORPO" versus placebo and versus untreated control area. Study products were applied once, on experimentally induced erythema by repeated tape stripping on 4 different adjacent skin areas of the forearms (volar surface - 2 areas on each side)
  Interventions: Other: P926 - LICHTENA DermAD CREMA VISO; Other: P927 - LICHTENA DermAD CREMA CORPO; Other: P926 - LICHTENA DermAD CREMA VISO - PLACEBO; Other: Untreated control area

INTERVENTIONS:
Other: P926 - LICHTENA DermAD CREMA VISO — The study product was applied on a skin areas of about 14 cm2 of the forearm, defined turning on the right and left side in accordance with a randomization list, on which an erythema has been experimentally induced by repeated tape stripping.
Other: P927 - LICHTENA DermAD CREMA CORPO — The study product was applied on a skin areas of about 14 cm2 of the forearm, defined turning on the right and left side in accordance with a randomization list, on which an erythema has been experimentally induced by repeated tape stripping.
Other: P926 - LICHTENA DermAD CREMA VISO - PLACEBO — The study product was applied on a skin areas of about 14 cm2 of the forearm, defined turning on the right and left side in accordance with a randomization list, on which an erythema has been experimentally induced by repeated tape stripping.
Other: Untreated control area — Untreated skin area of about 14 cm2 of the forearm, defined turning on the right and left side in accordance with a randomization list, on which an erythema has been experimentally induced by repeated tape stripping.

SUMMARY:
Open clinical study to evaluate the soothing and re-epithelizing activity of a single application of two cometic formulations ("P926 - LICHTENA DermAD CREMA VISO" and "P927 - LICHTENA DermAD CREMA CORPO") on experimentally induced erythema by repeated tape stripping on the forearm (volar surface) of 20 healthy volunteers.

Study products activity was assessed in comparison to placebo ("P926P - LICHTENA DermAD CREMA VISO - PLACEBO") and versus untreated control area.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers of both sexes
* TEWL value on tested skin areas immediately after tape stripping >15g/m2-h
* volunteers in a good general state of health in the Investigator opinion
* volunteers not taking drugs or undergoing surgical procedure
* volunteers who are giving a written informed consent.

Exclusion Criteria:

* Pregnancy (only for female subjects)
* lactation (only for female subjects)
* TEWL value on tested skin areas immediately after tape stripping <15g/m2-h
* change in the normal habits in the last month
* participation in a similar study during the previous month
* known allergy to one or several ingredients of the products on trial.
* Dermatitis
* presence of cutaneous disease on the tested area, as lesions, scars, malformations
* clinical and significant skin condition on the test area.
* Diabetes
* endocrine disease
* hepatic disorder
* renal disorder
* cardiac disorder
* pulmonary disease
* cancer
* neurological or psychological disease
* inflammatory/immunosuppressive disease
* drug allergy.
* Anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment starting more than 1 year ago);
* using of drugs able to influence the test results in the investigator opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline of skin erythema index | Baseline (T0), 1 hour (T1h), 24 hours (T24h)
  The instrumental measurement of erythema is performed by the use of an optical densitometer (X-RITE 404)
Change from baseline of skin redness | Baseline (T0), 1 hour (T1h), 24 hours (T24h)
  The instrumental measurement of skin redness is performed by the use of an optical colorimetry (Chroma Meter CR-200®)
Change from baseline of Transepidermal water loss (TEWL) | Baseline (T0), 1 hour (T1h), 24 hours (T24h)
  The measurement of TEWL, performed by the use of Tewameter® TM300, allows to objectively monitor skin responses to cosmetic treatments. A shift from low-normal rates of TEWL to high levels is due to barrier disruption.
Change from baseline of Superficial skin hydration | Baseline (T0), 1 hour (T1h), 24 hours (T24h)
  Skin electrical capacitance value is measured with Corneometer CM825
Change from baseline of deep skin hydration | Baseline (T0), 1 hour (T1h), 24 hours (T24h)
  Tissue dielectric constant of deep skin layers is measured with MoistureMeterD
Change from baseline of Epicutaneous pH | Baseline (T0), 1 hour (T1h), 24 hours (T24h)
  Surface cutaneous pH is measured with pH meter HI5221
Change from baseline of Surface microrelief's regularity | Baseline (T0), 1 hour (T1h), 24 hours (T24h)
  Surface microrelief's regularity is performed on skin replicas images acquired by Primos compact portable

CONTACTS AND LOCATIONS:
Locations (1):
- DERMING, Milan, MI, Italy